CLINICAL TRIAL: NCT03932799
Title: The Washington and Ohio Worker (WOW) Study: Comparing State Payer Strategies to Prevent Unsafe Opioid Prescribing
Brief Title: Comparing State Payer Strategies to Prevent Unsafe Opioid Prescribing
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Gary Franklin, Research Professor, School of Public Health: Environmental & Occupational Health, University of Washington
Other Study IDs: STUDY00006455; PCORI-UOP-2017C2-8509 (Other: PCORI)
Record Dates: First submitted 2019-04-19; First posted 2019-05-01 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Opioid Use; Opioid-Related Disorders
Keywords: Workers' Compensation; Occupational Injuries; Drug Utilization Review; Humans; Adult; Cohort Studies; Qualitative Research
MeSH Terms: conditions — Opioid-Related Disorders; Occupational Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Washington: Workers in the Washington Department of Labor and Industries state fund insurance system.
  Interventions: Other: Prospective prior authorization (PA) with hard stops in Washington
- Ohio: Workers in the Ohio Bureau of Workers' Compensation state fund insurance system.
  Interventions: Other: Retrospective review (RR) with prescriber notification in Ohio

INTERVENTIONS:
Other: Prospective prior authorization (PA) with hard stops in Washington — Under Washington regulatory procedures, payment for any opioid prescription billed beyond six weeks after the injury is denied unless the prescriber has submitted a checklist attesting to completion of all best practices from the regulations/guidelines.Thus, the Washington intervention is prospective and includes a "hard stop" subject to an insurer's decision based on regulatory authority.
  Groups: Washington
Other: Retrospective review (RR) with prescriber notification in Ohio — In Ohio an automated report identifies new opioid prescriptions beyond the acute phase. Ohio Workers' Compensation pharmacy and clinical staff review the medical record at 12 weeks to determine whether best practices were met. If not, the prescriber is notified via letter, and cases are reviewed again at 16 weeks. If best practices have still not been met, the prescriber and worker are notified via letter that opioid coverage will end in 4 weeks. The Ohio program relies on retrospective chart review and communication of best practices to prescribers.
  Groups: Ohio

SUMMARY:
This study examines the comparative effectiveness of opioid review programs in reducing unsafe opioid prescribing in two states: prospective prior authorization (PA) with hard stops in Washington and retrospective review (RR) with prescriber notification in Ohio.

DETAILED DESCRIPTION:
Use and misuse of opioids is now recognized as a major U.S. public health problem, leading to significant morbidity and mortality. Prescribing of both opioids and concurrent sedative-hypnotics for acute and chronic musculoskeletal pain increased dramatically from 2001 to 2010. The clearest path to preventing transition to chronic opioid use and associated morbidity or addiction is to reduce unnecessary prescribing during the acute (0-6 weeks) and subacute (6-12 weeks) phases of pain.

Both prior authorization (PA) and other insurer-based drug utilization programs are increasingly being used in an attempt to stem the tide of the opioid epidemic and to reduce unsafe opioid prescribing. Review programs have proven effective in decreasing use and overall costs of more expensive medications. Washington (WA) and Ohio (OH) offer a unique opportunity to study opioid prescribing interventions because both states have regulatory authority over health care delivery to all injured workers, and are the two largest states with a population-based exclusive State Fund. Further, both states have initiated distinct prescribing guideline-concordant opioid review programs (ORPs), allowing for a unique natural experiment to compare the effectiveness of two substantially different approaches to reducing unsafe opioid prescribing.

This is an observational cohort study, with prospective and retrospective components. Aims 1 and 2 rely primarily on administrative data for a prospective cohort, with longitudinal surveys conducted among a subset of the cohort. Aim 1 also includes a retrospective time series analysis. Aim 3 relies on qualitative research, including individual in-depth interviews and key informant interviews.

Specific aim 1. Examine the comparative effectiveness of prospective prior authorization (PA) with hard stops in WA versus retrospective review (RR) with prescriber notification in OH in reducing unsafe opioid prescribing.

Specific aim 2. Examine the comparative effectiveness of WA's PA program versus OH's RR program with regard to patient reported outcomes (pain, function, quality of life, return to work), harms (presence of opioid use disorder, opioid poisoning events) and work disability outcomes at 6 weeks, 6 months, and 12 months from date of injury.

Specific aim 2a. For injured workers in WA, examine unsafe opioid prescribing and patient-reported outcomes and work disability at 6 and 12 months for patients receiving an established, coordinated, stepped care management program during the first 12 weeks following injury plus prospective PA versus patients receiving usual care subject to PA only.

Specific aim 3. Using qualitative methods, identify key environmental, programmatic and policy factors that influenced the design, implementation and impact of the PA program in WA and the RR program in OH. This information will lead to the development of an Opioid Review Tool educational module for dissemination to both public and private payers.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2:

* File a new accepted State Fund claim
* Fill at least one opioid prescription, paid for by workers' compensation, during the first 6 weeks after date of injury

Aim 3 key informants

* Policy makers and stakeholders who were involved in the creation and implementation of the Washington or Ohio opioid review program.

Aim 3 individual in-depth interviews

* Providers that had at least one patient whose opioid prescriptions paid for through workers' compensation had been reviewed in accordance with the state's opioid review program.
* Patients that had an opioid prescription for at least 6 weeks paid for by workers' compensation or whose prescription payments have been reviewed in accordance with the state's opioid review program.

Exclusion Criteria (Aims 1 and 2):

* Under 18 years of age
* Current cancer diagnosis
* Surveys only: do not speak English or Spanish, physically or mentally incapable of completing the survey, incarcerated, deceased

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Workers in the Washington Department of Labor and Industries or Ohio Bureau of Workers' Compensation state fund insurance system.
Sampling Method: Non-Probability Sample
Enrollment: 5411 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Franklin, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Washington: Injured workers in the Washington Department of Labor and Industries (L&I) state fund insurance system - required to obtain prior authorization for opioids prescribed after 6 weeks from an injury.
- Ohio: Injured workers in the Ohio Bureau of Workers' Compensation (BWC) state fund insurance system - subject to a retrospective review of claim if receiving opioid prescription after 6 weeks from injury. Prescriber notified if best practices are not being documented.
Period: Overall Study
Arm/Group | Washington | Ohio
Started | 4632 | 779
Completed | 4632 | 779
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Washington | Ohio | Total
Number analyzed (Participants) | 4632 | 779 | 5411
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 440 | 51 | 491
  25-34 | 1100 | 167 | 1267
  35-44 | 1121 | 154 | 1275
  45-54 | 1033 | 175 | 1208
  55-64 | 791 | 187 | 978
  ≥65 | 147 | 45 | 192
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 17 participants in Ohio missing data on sex.
  Participants
    number analyzed (Participants) | 4632 | 762 | 5394
    Female | 1153 | 193 | 1346
    Male | 3479 | 569 | 4048
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subacute Phase - More Than 7 Days of Opioids
Description: More than 7 unique days of opioids within the time period
Time Frame: 6-12 weeks after injury
Measure: Number; unit: % of participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 4632 | 779
% of participants | 1.9 | 12.2
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Robust variance estimates; Test type: Superiority — Adjusted for workers' compensation-based covariates: age, gender, urban/rural residence, coronavirus disease (COVID)-19 era injury, days from injury to Report of Accident, injury type, injury complexity/severity, days from injury to first opioid prescription, more than 7 days of opioids in acute phase, and health care utilization during baseline period/acute phase; p < .001, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.16 to 0.38]

2. Primary Outcome: Chronic Phase - Composite (Meeting ≥1 of the 3 Chronic Phase Metrics)
Description: At least 1 instance of either chronic opioid prescribing, concurrent opioid and sedative prescribing, or high dose opioid prescribing attributed to a worker within the time period
Time Frame: 3-6, 6-9, and 9-12 months after injury
Measure: Number; unit: % of participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 4632 | 779
% of participants
  3-6 months | 1.2 | 2.4
  6-9 months | 0.9 | 2.4
  9-12 months | 0.8 | 2.1
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Outcome modeled longitudinally over the 3 time periods (3-6, 6-9, and 9-12 months) * Time periods clustered at the individual worker level * Exchangeable working correlation structure * Robust variance estimates; Test type: Superiority — Adjusted for workers' compensation-based covariates: age, gender, urban/rural residence, COVID-19 era injury, days from injury to Report of Accident, injury type, injury complexity/severity, days from injury to first opioid prescription, more than 7 days of opioids in acute phase, health care utilization during baseline period/acute phase, and time indicator for each time period (0,1,2); p = .43, Generalized estimating equation — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.53 to 1.31]

3. Primary Outcome: Chronic Phase - Chronic Opioids (≥60 Days' Supply)
Description: 60 or more unique days of opioids within the time period
Time Frame: 3-6, 6-9, and 9-12 months after injury
Measure: Number; unit: % of participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 4632 | 779
% of participants
  3-6 months | 0.0 | 1.7
  6-9 months | 0.0 | 2.3
  9-12 months | 0.0 | 1.9

4. Primary Outcome: Chronic Phase - Concurrent (Concurrent Sedatives/Hypnotics and Opioids on ≥1 Day)
Description: At least 1 overlapping day of both a sedative and an opioid within the time period
Time Frame: 3-6, 6-9, and 9-12 months
Measure: Number; unit: % of participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 4632 | 779
% of participants
  3-6 months | 0.0 | 0.4
  6-9 months | 0.0 | 0.1
  9-12 months | 0.0 | 0.1

5. Primary Outcome: Chronic Phase - High Dose (Average of ≥50 Morphine Equivalent Daily Dose [MEDD] Among All Days With Opioids)
Description: Mean MEDD of 50 or more during the days a worker received opioids (based on days' supply) within the time period
Time Frame: 3-6, 6-9, and 9-12 months after injury
Measure: Number; unit: % of participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 4632 | 779
% of participants
  3-6 months | 1.2 | 1.0
  6-9 months | 0.9 | 0.5
  9-12 months | 0.8 | 0.4
Statistical Analysis 1: Comparison: Washington vs Ohio; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .002, Generalized estimating equation — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.50 to 6.14]

6. Secondary Outcome: ≥30% Decrease in Pain Intensity/Interference (PEG-3)
Description: Clinically important improvement in pain intensity/interference defined as obtaining a ≥30% reduction in pain intensity and interference from baseline. This was assessed with the PEG-3, which is comprised of 3 items assessing pain intensity and pain interference with enjoyment of life/general activity on a 0 to 10 numerical rating scale (0 = no pain/does not interfere, 10 = pain as bad as you can imagine/completely interferes).
  1 = ≥30% reduction in mean PEG-3 summary score from baseline; 0 = otherwise.
Time Frame: 12 months after injury
Population: * Analysis performed within a distinct survey sample of workers
  * Estimates for Washington (WA) have been survey-weighted; sampling weights for Ohio (OH) were always 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 1001 | 151
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — Adjusted for same covariates as primary outcomes, plus survey covariates: days from injury to baseline survey, education, household income, race/ethnicity, working for pay, recovery expectations, anxious symptoms, depressive symptoms, pre-injury opioid, chiropractic and physical therapy (PT) utilization during baseline period/acute phase, cannabis for injury pain, alcohol misuse risk, current tobacco use, pain intensity/interference, Functional Comorbidity Index, health status, quality of life; p = .84, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.71 to 1.32]

7. Secondary Outcome: Anxious Symptoms (PHQ-4)
Description: 2-item PHQ-4 subscale assessed how often participant was bothered by anxious symptoms on 4-point scale (0 = not at all, 3 = nearly every day).
  1 = summed subscale score ≥3; 0 = otherwise.
Time Frame: 12 months after injury
Population: * Analysis performed within a distinct survey sample of workers
  * Estimates for WA have been survey-weighted; sampling weights for OH were always 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 487 | 79
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — Adjusted for same covariates as primary outcomes, plus survey-based covariates: days from injury to baseline survey date, education, household income, race/ethnicity, working for pay, recovery expectations, anxious symptoms, depressive symptoms, pre-injury opioid, chiropractic and PT utilization during baseline period/acute phase, cannabis for injury pain, alcohol misuse risk, current tobacco use, pain intensity/interference, Functional Comorbidity Index, health status, and quality of life; p = .88, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.71 to 1.49]

8. Secondary Outcome: Depressive Symptoms (PHQ-4)
Description: 2-item PHQ-4 subscale assessing how often participant was bothered by depressive symptoms on 4-point scale (0 = not at all, 3 = nearly every day).
  1 = summed subscale score ≥3; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 322 | 64
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .15, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.49 to 1.11]

9. Secondary Outcome: Global Improvement (GIC)
Description: Global Impression of Change on 7-point Likert scale. Participants asked to rate how they compared now to immediately after their injury (1 = very much improved, 7 = very much worse)
  1 = "much improved" or "very much improved"; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 1413 | 222
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .38, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.60 to 1.21]

10. Secondary Outcome: Disability - Activity Limitation
Description: Modified activity limitation items from the National Health Interview Survey (NHIS) 2011 Adult Functioning Supplement. Participants were asked to rate on a 3-point scale (limited a lot, limited a little, not limited at all) whether their health was limited in four domains: participating in leisure or social activities, getting out with friends or family, doing household chores such as cooking and cleaning, and using transportation to get to places you want to go.
  1 = "limited a lot" ; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants
  Leisure or social activities | 281 | 49
  Getting out with friends or family | 220 | 37
  Doing household chores | 246 | 56
  Using transportation | 137 | 22
Statistical Analysis 1: Comparison: Washington vs Ohio; * Leisure or social activities outcome * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .12, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.91 to 2.28]
Statistical Analysis 2: Comparison: Washington vs Ohio; * Getting out with friends or family outcome * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .42, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.74 to 2.07]
Statistical Analysis 3: Comparison: Washington vs Ohio; * Doing household chores outcome * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .91, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.63 to 1.51]
Statistical Analysis 4: Comparison: Washington vs Ohio; * Using transportation outcome * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .59, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.64 to 2.21]

11. Secondary Outcome: Not Working for Pay
Description: Participants asked whether they worked for pay in the past week.
  1 = did not work for pay in the week prior to assessment; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 599 | 107
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .22, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.88 to 1.75]

12. Secondary Outcome: On Time Loss (Not Working)
Description: 1 = on time loss (workers' compensation warrant data); 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 209 | 43
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .02, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.12 to 3.47]

13. Secondary Outcome: Earning Less Than Before Injury
Description: Participants asked to rate on a 5-point Likert scale the extent to which earnings differed from earnings at time of injury (1 = a lot more than before the injury, 5 = a lot less than before the injury).
  1 = "somewhat less than before", "a lot less than before the injury", or not working; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 819 | 129
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .10, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.95 to 1.83]

14. Secondary Outcome: Opioid Overdose/Adverse Effects
Description: Qualifying International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnosis codes: first 3 digits = "T40" and 5th digit = ("0","1","2","3","4","6") and 7th digit not = "6" (excludes underdosing).
  1 = presence of qualifying ICD-10-CM diagnosis code; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 2 | 0

15. Secondary Outcome: Quality of Life (EuroQol EQ-5D)
Description: 5-item scale in which participants were asked to rate the extent to which they experienced problems with mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale (1 = no problems, 5 = extreme problems). Individual item responses were used to create score profiles (range 11111 to 55555), which were then converted to an index value using a US-based value set.
  -0.573 (worst health state) to 1 (best health state)
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: index value
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
index value | 0.81 (0.16) | 0.79 (0.16)
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .53, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; beta = -0.01, 95% CI 2-sided [-0.03 to 0.01]

16. Secondary Outcome: Satisfaction With Overall Treatment
Description: Single-item 5-point Likert scale rating of how satisfied participants were with all injury-related treatment (-2 = very dissatisfied, 2 = very satisfied).
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on 5-point Likert scale
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
score on 5-point Likert scale | 0.98 (1.17) | 0.81 (1.32)
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .053, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; beta = 0.16, 95% CI 2-sided [-0.00 to 0.32]

17. Secondary Outcome: Satisfaction With Pain-related Treatment
Description: Single-item 5-point Likert scale rating of how satisfied participants were with treatment received for injury-related pain (-2 = very dissatisfied, 2 = very satisfied).
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on 5-point Likert scale
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
score on 5-point Likert scale | 0.88 (1.26) | 0.66 (1.34)
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .01, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; beta = 0.22, 95% CI 2-sided [0.05 to 0.38]

18. Other Pre Specified Outcome: Problematic Opioid Use (TAPS)
Description: 3-item TAPS tool Part 2 assessing any problematic opioid use in the past 3 months. Participants asked if they used a prescription opioid not as prescribed, if they failed in cutting down on opioid use, and if anyone has expressed concern about their opioid use (0 = no, 1 = yes). The items were summed to create a summary score in which scores ≥1 represented problematic or high-risk opioid use.
  1 = summed subscale score ≥1; 0 = otherwise.
Time Frame: 12 months after injury
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Washington | Ohio
Number analyzed (Participants) | 1976 | 319
Participants | 113 | 22
Statistical Analysis 1: Comparison: Washington vs Ohio; * Primary predictor is binary (1 for Washington, 0 for Ohio) * Models survey weighted * Robust variance estimates; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = .35, Regression, Logistic — * two-tailed test * p-values < 0.05 are statistically significant; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.42 to 1.35]

ADVERSE EVENTS:
Description: Adverse event data were not collected for this observational study.
Arm/Group | Washington | Ohio
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03932799/Prot_SAP_000.pdf